CLINICAL TRIAL: NCT00602771
Title: A Randomized Phase II Trial of Tipifarnib (R115777, ZARNESTRA, NSC #702818) in Combination With Oral Etoposide (VP-16) in Elderly Adults With Newly Diagnosed, Previously Untreated Acute Myelogenous Leukemia (AML)
Brief Title: Tipifarnib and Etoposide in Treating Older Patients With Newly Diagnosed, Previously Untreated Acute Myeloid Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00278; NCI-2009-00278 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000584212; J07109 (Other: Johns Hopkins University/Sidney Kimmel Cancer Center); 8077 (Other: CTEP); N01CM62204 (NIH); P30CA006973 (NIH); U01CA070095 (NIH)
Record Dates: First submitted 2008-01-19; First posted 2008-01-28 (Estimated); Results first posted 2014-05-26 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-06

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Secondary Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute; Leukemia, Erythroblastic, Acute | interventions — tipifarnib; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Experimental): Patients receive 600 mg of oral tipifarnib twice daily on days 1-14 and 100 mg of oral etoposide once daily on days 1-3 and 8-10.
  Interventions: Drug: tipifarnib; Drug: etoposide
- Arm II (closed to accrual as of November 2008) (Experimental): Patients receive 400 mg of oral tipifarnib twice daily on days 1-14 and 200 mg of oral etoposide once daily on days 1-3 and 8-10.
  Interventions: Drug: tipifarnib; Drug: etoposide

INTERVENTIONS:
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra
Drug: etoposide — Given orally
  Other Names: EPEG; VP-16; VP-16-213

SUMMARY:
This randomized phase II trial is studying the side effects and how well giving tipifarnib together with etoposide works in treating older patients with newly diagnosed, previously untreated acute myeloid leukemia. Tipifarnib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as etoposide, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Giving tipifarnib together with etoposide may kill more cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. To compare the efficacy and toxicity of two schedules of tipifarnib plus etoposide as induction therapy in older patients with newly diagnosed, previously untreated acute myeloid leukemia.

II. To study mechanisms of leukemia cell resistance to tipifarnib in combination with etoposide.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive 600 mg of oral tipifarnib twice daily on days 1-14 and 100 mg of oral etoposide once daily on days 1-3 and 8-10.

ARM II: Patients receive 400 mg of oral tipifarnib twice daily on days 1-14 and 200 mg of oral etoposide once daily on days 1-3 and 8-10. (closed to accrual as of November 2008)

Treatment in both arms repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 30 days and then every 90 days thereafter.

ELIGIBILITY:
Criteria:

* Pathologically confirmed newly diagnosed acute myeloid leukemia (AML)
* Subtypes M0, M1, M2, M4-7 disease
* No newly diagnosed acute promyelocytic leukemia (M3)
* Any of the following diseases:
* De novo disease
* Secondary AML
* Myelodysplasia (MDS)-related AML (MDS/AML)
* Treatment-related AML
* Previously untreated disease
* Patients who have received prior hydroxyurea alone or non-cytotoxic therapies for MDS (e.g., thalidomide, interferon, cytokines, 5-azacytidine, or revlimid) will be eligible for this study
* Must be considered ineligible for traditional antileukemia chemotherapy
* No hyperleukocytosis with ≥ 30,000 blasts/uL or rapidly rising blast count with projected doubling time of =< 2 days
* Patients may receive hydroxyurea to lower blast count to < 30,000 blasts/uL up to 24 hours before beginning tipifarnib and etoposide
* No active CNS leukemia
* No prior tipifarnib or etoposide
* No concurrent radiotherapy, immunotherapy, or other chemotherapy
* No concurrent enzyme-inducing anticonvulsants (e.g., phenytoin, fosphenytoin, phenobarbital, primidone, carbamazepine, or oxcarbazepine)
* Patients may be changed to non-enzyme-inducing anticonvulsants and stabilized before starting study treatment

Inclusion Criteria:

* ECOG performance status 0-2
* Serum creatinine =< 2.0 mg/dL
* SGOT and SGPT =< 3 times upper limit of normal
* Bilirubin =< 2 mg/dL

Exclusion Criteria:

* Active, uncontrolled infection
* Patients with infection under active treatment and controlled with antimicrobials are eligible
* Presence of other life-threatening illnesses
* Patients with mental deficits and/or psychiatric history that preclude them from giving informed consent or from following protocol
* Allergies to imidazoles (e.g., clotrimazole, ketoconazole, miconazole, or econazole)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 84 (Actual)
Dates: Start 2008-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Judith Karp, Principal Investigator — Johns Hopkins University/Sidney Kimmel Cancer Center
Locations (5):
- United States (5):
  - Blood and Marrow Transplant Group of Georgia, Atlanta, Georgia
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Weill Medical College of Cornell University, New York, New York

REFERENCES:
- [Derived] Ding H, McDonald JS, Yun S, Schneider PA, Peterson KL, Flatten KS, Loegering DA, Oberg AL, Riska SM, Huang S, Sinicrope FA, Adjei AA, Karp JE, Meng XW, Kaufmann SH. Farnesyltransferase inhibitor tipifarnib inhibits Rheb prenylation and stabilizes Bax in acute myelogenous leukemia cells. Haematologica. 2014 Jan;99(1):60-9. doi: 10.3324/haematol.2013.087734. Epub 2013 Aug 30. PMID 23996484
- [Derived] Karp JE, Vener TI, Raponi M, Ritchie EK, Smith BD, Gore SD, Morris LE, Feldman EJ, Greer JM, Malek S, Carraway HE, Ironside V, Galkin S, Levis MJ, McDevitt MA, Roboz GR, Gocke CD, Derecho C, Palma J, Wang Y, Kaufmann SH, Wright JJ, Garret-Mayer E. Multi-institutional phase 2 clinical and pharmacogenomic trial of tipifarnib plus etoposide for elderly adults with newly diagnosed acute myelogenous leukemia. Blood. 2012 Jan 5;119(1):55-63. doi: 10.1182/blood-2011-08-370825. Epub 2011 Oct 14. PMID 22001391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: January 2008 and December 2009,
Pre-assignment Details: 5 patients signed consent, but were deemed screen failures and did not begin study treatment
Period: Overall Study
Arm/Group | Arm I | Arm II (Closed to Accrual as of November 2008)
Started | 63 | 21
Completed | 62 | 21
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I | Arm II (Closed to Accrual as of November 2008) | Total
Number analyzed (Participants) | 63 | 21 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 63 | 21 | 84
Age, Continuous [Mean (Standard Deviation); unit: years] | 76 (20) | 78 (19) | 76 (20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 7 | 31
  Male | 39 | 14 | 53
Region of Enrollment [Number; unit: participants]
  United States | 63 | 21 | 84

OUTCOME MEASURES:

1. Primary Outcome: Complete Response
Description: Bone marrow showing less than 5% myeloblasts with normal maturation of all cell lines, an ANC of at least 1000/mcL and a platelet count of 100,000 mcL, absence of blast in peripheral blood, absence of identifiable leukemic cells in the bone marrow, clearance of disease-associated cytogenetic abnormalities, and clearance of any previously existing extramedullary disease. A CR must be confirmed 4 to 6 weeks after the initial documentation. If possible, at least one bone marrow biopsy should be performed to confirm the CR.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Arm I | Arm II (Closed to Accrual as of November 2008)
Number analyzed (Participants) | 15 | 6
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm I | Arm II (Closed to Accrual as of November 2008)
Serious Adverse Events (participants affected / at risk) | 5/63 | 8/21
Other Adverse Events (participants affected / at risk) | 18/63 | 6/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=63) | Arm II (Closed to Accrual as of November 2008) (N=21)
non-hematologic toxicities (General disorders) | 4 (4) | 7 (7) — All grade 3 non-hematologic toxicities from table 2 of the manuscript
Infections (Infections and infestations) | 5 (5) | 8 (8) — Grade 3 or greater
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (N=63) | Arm II (Closed to Accrual as of November 2008) (N=21)
Dose reduction (Nervous system disorders) | 18 (18) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less